CLINICAL TRIAL: NCT05113940
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, SPONSOR-OPEN, PLACEBO-CONTROLLED STUDY TO INVESTIGATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS, AND PHARMACOKINETIC INTERACTION WITH MIDAZOLAM OF MULTIPLE ASCENDING ORAL DOSES OF PF-07258669 IN HEALTHY NON-JAPANESE AND JAPANESE ADULT PARTICIPANTS
Brief Title: A Study of PF-07258669 In Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: C4541003; 2021-004037-36 (EudraCT Number)
Record Dates: First submitted 2021-10-13; First posted 2021-11-09 (Actual); Results first posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-07

CONDITIONS: Healthy Participants
Keywords: PF-07258669; multiple dose; melanocortin-4 receptor; MC4R; healthy participants; safety; tolerability; pharmacokinetics
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (13):
- PF-07258669 and Placebo (Cohort 1) (Experimental): Dose level 1: Multiple dose administration of PF-07258669 and placebo over 14 days in non-Japanese participants; 8 participants will receive PF-07258669 and 2 will receive placebo Dietary allocation: High Carbohydrate High Calorie (HCHC)
  Interventions: Drug: PF-07258669; Drug: Placebo
- PF-07258669 and Placebo (Cohort 2) (Experimental): Dose level 2: Multiple dose administration of PF-07258669 and placebo over 14 days in non-Japanese participants; 8 participants will receive PF-07258669 and 2 will receive placebo Dietary allocation: HCHC
  Interventions: Drug: PF-07258669; Drug: Placebo
- PF-07258669 and Placebo (Cohort 3) (Experimental): Dose level 3: Multiple dose administration of PF-07258669 and placebo over 14 days in non-Japanese participants; 8 participants will receive PF-07258669 and 2 will receive placebo Dietary allocation: HCHC
  Interventions: Drug: PF-07258669; Drug: Placebo
- PF-07258669 and Placebo (Cohort 4) (Experimental): Dose level 4: Multiple dose administration of PF-07258669 and placebo over 14 days in non-Japanese participants; 8 participants will receive PF-07258669 and 2 will receive placebo Dietary allocation: Standard Diet (SD)
  Interventions: Drug: PF-07258669; Drug: Placebo
- PF-07258669 and Placebo (Cohort 5) (Experimental): Dose level 5: Multiple dose administration of PF-07258669 and placebo over 14 days in non-Japanese participants; 8 participants will receive PF-07258669 and 2 will receive placebo Dietary allocation: SD
  Interventions: Drug: PF-07258669; Drug: Placebo
- PF-07258669 and Placebo (Cohort 6) (Experimental): Multiple dose administration of PF-07258669 and placebo over 14 days in Japanese participants; 8 participants will receive PF-07258669 and 2 will receive placebo Dietary allocation: SD
  Interventions: Drug: PF-07258669; Drug: Placebo
- Midazolam with and without PF-07258669 (Cohort 8) (Experimental): Drug-drug interaction assessment of pharmacokinetics interaction in PF-07258669 and midazolam Dietary allocation: SD
  Interventions: Drug: PF-07258669; Drug: Midazolam
- PF-07258669 and Placebo (Cohort 7) (Experimental): Multiple dose administration of PF-07258669 and placebo over 14 days in older adult participants; 8 participants will receive PF-07258669 and 2 will receive placebo Dietary allocation: SD
  Interventions: Drug: PF-07258669; Drug: Placebo
- PF-07258669 and Placebo (Cohort 9) (Experimental): Dose level 6: Multiple dose administration of PF-07258669 and placebo over 14 days in non-Japanese participants; 8 participants will receive PF-07258669 and 2 will receive placebo Dietary allocation: SD
  Interventions: Drug: PF-07258669; Drug: Placebo
- PF-07258669 and Placebo (Cohort 10) (Experimental): Dose level 7: Multiple dose administration of PF-07258669 and placebo over 14 days in non-Japanese participants; 8 participants will receive PF-07258669 and 2 will receive placebo Dietary allocation: SD
  Interventions: Drug: PF-07258669; Drug: Placebo
- PF-07258669 and Placebo (Cohort 11) (Experimental): Dose level 8: Multiple dose administration of PF-07258669 and placebo over 14 days in non-Japanese participants; 8 participants will receive PF-07258669 and 2 will receive placebo Dietary allocation: SD
  Interventions: Drug: PF-07258669; Drug: Placebo
- PF-07258669 and Placebo (Cohort 12) (Experimental): Dose Level 9: Multiple dose administration of PF-07258669 and placebo over 14 days in non-Japanese participants; 8 participants will receive PF-07258669 and 2 will receive placebo Dietary allocation: High Fat High Calorie (HFHC)
  Interventions: Drug: PF-07258669; Drug: Placebo
- PF-07258669 and Placebo (Cohort 13) (Experimental): Dose Level 10: Multiple dose administration of PF-07258669 and placebo over 14 days in non-Japanese participants; 8 participants will receive PF-07258669 and 2 will receive placebo Dietary allocation: High Fat High Calorie (HFHC)
  Interventions: Drug: PF-07258669; Drug: Placebo

INTERVENTIONS:
Drug: PF-07258669 — PF-07258669 will be administered as tablets; every 8 hour (Q8H) or every 12 hour (Q12H) over 14 days
Drug: Placebo — Placebo will be administered as tablets; Q8H or Q12H over 14 days
  Arms: PF-07258669 and Placebo (Cohort 1); PF-07258669 and Placebo (Cohort 10); PF-07258669 and Placebo (Cohort 11); PF-07258669 and Placebo (Cohort 12); PF-07258669 and Placebo (Cohort 13); PF-07258669 and Placebo (Cohort 2); PF-07258669 and Placebo (Cohort 3); PF-07258669 and Placebo (Cohort 4); PF-07258669 and Placebo (Cohort 5); PF-07258669 and Placebo (Cohort 6); PF-07258669 and Placebo (Cohort 7); PF-07258669 and Placebo (Cohort 9)
Drug: Midazolam — Single doses of Midazolam will be administered as oral solution alone and in combination with PF-07258669
  Arms: Midazolam with and without PF-07258669 (Cohort 8)

SUMMARY:
Part A of this study is to evaluate safety, tolerability, and pharmacokinetics (PK) of PF-07258669 after administration of multiple ascending oral doses to healthy adult participants. Optional cohorts of healthy adult Japanese participants and/or older adult participants may also be evaluated if results in other cohorts support further evaluation. Part B of this study is a 2-period, fixed-sequence, multiple-dose, open-label design to evaluate the effect of PF-07258669 on midazolam PK in healthy adult participants. Part B will be conducted if the results of Part A support further evaluation of PF-07258669.

ELIGIBILITY:
Inclusion Criteria:

1. For optional cohort of older adult participants only: Male participants and female participants of non childbearing potential must be 65 to 90 years of age, inclusive, at the time of signing the ICD (informed consent document). Attempts will be made to ensure that the age composition of this cohort (eg, approximately 70% of participants ≥70 years of age) is comparable to that of the anticipated patient population in later clinical studies.
2. Female participants of nonchildbearing potential and male participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.

   For optional cohort of older adult participants only: Participants must be in a stable condition at admission. These participants must be in reasonably good health as determined by the investigator based on a detailed medical history, full physical examination, vital signs assessments, 12-lead ECG (electrocardiogram), and clinical laboratory tests. Participants with mild, chronic, stable disease (eg, controlled hypertension, noninsulin dependent diabetes, osteoarthritis) may be enrolled if deemed medically prudent by the investigator.
3. Participants who are willing to avoid direct sunlight exposure or any high intensity ultraviolet light exposure from admission to the follow-up contact and to apply sunscreen/lotion with a high sun protection factor and to wear eye protection, as appropriate.
4. Body mass index (BMI) of 17.5 to 28.5 kg/m2; and a total body weight >50 kg (110 lb).

   For optional cohort of older adult participants only: BMI of 17.5 to 32.4 kg/m2; and a total body weight >50 kg (110 lbs). Efforts will be made to enroll at least 3 older adult participants with BMI <25 kg/m2, if feasible.
5. Japanese participants only: Participants enrolling as Japanese must have 4 biological Japanese grandparents who were born in Japan.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine (including, but not limited to, thyroid disease, diabetes insipidus), pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric (including, but not limited to, primary polydipsia, obsessive compulsive disorder, anxiety disorder, schizophrenia), neurological (including, but not limited to, seizure disorder, traumatic brain injury), immunodeficiency (including, but not limited to, severe infection that required ICU admission, prolonged hospitalization, or prolonged treatment) or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing), as well as presence of clinical laboratory abnormalities.

   For optional cohort of older adult participants only: Participants with chronic conditions (eg, hypertension) that are controlled by either diet or stable doses of medications may be included. Recent evidence (ie, within previous 6 months) or history of unstable disease or moderate to severe conditions which would, in the investigator's opinion, interfere with the study evaluations or have an impact on the safety of participants.
2. History of symptomatic orthostatic hypotension or symptomatic bradycardia.
3. History of eating disorders (eg, anorexia or bulimia nervosa, binge-eating disorder, avoidant/restrictive food intake disorder).
4. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention.

   For optional cohort of older adult participants only: Participants taking daily prescription or non-prescription medications (that are not moderate or strong cytochrome P450 (CYP3A) inducers or inhibitors) for management of acceptable chronic medical conditions are to be on a stable dose, as defined by no change in dose for the 28 days or 5 half-lives (whichever is longer) before the screening visit.
   1. Use of stable concomitant mediations noted above that are CYP3A substrates may be restricted.
   2. All medications must be reviewed on a case-by-case basis by the investigator and approved by the sponsor during the screening period for eligibility purposes.
5. Use of moderate or strong cytochrome P450 3A (CYP3A) inhibitors or inducers within 28 days or 5 half-lives (whichever is longer) prior to first dose of study intervention.
6. Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).
7. Fasting serum triglycerides >2× ULN (upper limit of normal).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4541003

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consisted of two parts: Part A and Part B. A total of 120 participants were enrolled in the study.
Pre-assignment Details: Part A of this study was placebo-controlled evaluation of safety, tolerability, and PK of PF-07258669 after multiple ascending oral doses to healthy adult participants under 3 different dietary allocations: standard, high-carbohydrate high-calorie (HCHC), and high-fat, high-calorie (HFHC) diets. Part B was a 2-period, fixed-sequence, multiple-dose design to evaluate the effect of PF-07258669 on midazolam PK in healthy adult participants.
Groups:
- Placebo: 18-60 Years (HC-HC Diet): Healthy non-Japanese participants aged 18-60 years who were on high carbohydrate-high calorie (HC-HC) diet, received placebo matched to PF-07258669 tablets orally, every eight hours (Q8H) for 14 consecutive days (only a single morning dose administered on Day 14).
- PF-07258669 2 mg: 18-60 Years (HC-HC Diet): Healthy non-Japanese participants aged 18-60 years who were on HC-HC diet, received PF-07258669 2 milligrams (mg) tablets orally, Q8H for 14 consecutive days (only a single morning dose administered on Day 14).
- PF-07258669 3 mg: 18-60 Years (HC-HC Diet): Healthy non-Japanese participants aged 18-60 years who were on HC-HC diet, received oral PF-07258669 3 mg tablets orally, Q8H for 14 consecutive days (only a single morning dose administered on Day 14).
- PF-07258669 6 mg: 18-60 Years (HC-HC Diet): Healthy non-Japanese participants aged 18-60 years who were on HC-HC diet, received PF-07258669 6 mg tablets orally, Q8H for 14 consecutive days (only a single morning dose administered on Day 14).
- Placebo: 18-60 Years (Standard Diet): Healthy non-Japanese participants aged 18-60 years who were on standard diet, received placebo matched to PF-07258669 tablets orally, Q8H for 14 consecutive days (only a single morning dose administered on Day 14).
- PF-07258669 6 mg: 18-60 Years (Standard Diet): Healthy non-Japanese participants aged 18-60 years who were on standard diet, received PF-07258669 6 mg tablets orally, Q8H for 14 consecutive days (only a single morning dose administered on Day 14).
- PF-07258669 20 mg: 18-60 Years (Standard Diet): Healthy non-Japanese participants aged 18-60 years who were on standard diet, received PF-07258669 20 mg tablets orally, Q8H for 14 consecutive days (only a single morning dose administered on Day 14).
- PF-07258669 60 mg: 18-60 Years (Standard Diet): Healthy non-Japanese participants aged 18-60 years who were on standard diet, received PF-07258669 60 mg tablets orally, Q8H for 14 consecutive days (only a single morning dose administered on Day 14).
- PF-07258669 125 mg: 18-60 Years (Standard Diet): Healthy non-Japanese participants aged 18-60 years who were on standard diet, received PF-07258669 125 mg tablets orally, Q8H for 14 consecutive days (only a single morning dose administered on Day 14).
- PF-07258669 180 mg: 18-60 Years (Standard Diet): Healthy non-Japanese participants aged 18-60 years who were on standard diet, received PF-07258669 180 mg tablets orally, Q8H for 14 consecutive days (only a single morning dose administered on Day 14).
- Placebo: 18-60 Years (HF-HC Diet): Healthy participants aged 18-60 years who were on high fat-high calorie (HF-HC) diet, received placebo matched to PF-07258669 tablets orally, Q8H for 14 consecutive days (only a single morning dose administered on Day 14).
- PF-07258669 180 mg: 18-60 Years (HF-HC Diet): Healthy non-Japanese participants aged 18-60 years who were on HF-HC diet, received PF-07258669 180 mg tablets orally, Q8H for 14 consecutive days (only a single morning dose administered on Day 14).
- Placebo: Japanese 18-60 Years (Standard Diet): Healthy Japanese participants aged 18-60 years who were on standard diet, received placebo matched to PF-07258669 tablets orally, Q8H for 14 consecutive days (only a single morning dose administered on Day 14).
- PF-07258669 180 mg: Japanese 18-60 Years (Standard Diet): Healthy Japanese participants aged 18-60 years who were on standard diet, received PF-07258669 180 mg tablets orally, Q8H for 14 consecutive days (only a single morning dose administered on Day 14).
- Midazolam Then PF-07258669 + Midazolam: Standard Diet: Healthy non-Japanese participants aged 18-60 years who were on standard diet, received midazolam 1 milligram (mg) oral solution on Day 1 of Period 1 and then oral PF-07258669 180 mg tablets, Q8H from Day 1 to Day 10 of Period 2. On Days 2 and 10 of Period 2, participants received midazolam 1 mg oral solution.
Period: Part A (18 Days)
Arm/Group | Placebo: 18-60 Years (HC-HC Diet) | PF-07258669 2 mg: 18-60 Years (HC-HC Diet) | PF-07258669 3 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (HC-HC Diet) | Placebo: 18-60 Years (Standard Diet) | PF-07258669 6 mg: 18-60 Years (Standard Diet) | PF-07258669 20 mg: 18-60 Years (Standard Diet) | PF-07258669 60 mg: 18-60 Years (Standard Diet) | PF-07258669 125 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (Standard Diet) | Placebo: 18-60 Years (HF-HC Diet) | PF-07258669 180 mg: 18-60 Years (HF-HC Diet) | Placebo: Japanese 18-60 Years (Standard Diet) | PF-07258669 180 mg: Japanese 18-60 Years (Standard Diet) | Midazolam Then PF-07258669 + Midazolam: Standard Diet
Started | 6 | 8 | 8 | 7 | 10 | 8 | 8 | 8 | 8 | 8 | 12 | 12 | 1 | 5 | 0
Completed | 6 | 8 | 7 | 6 | 9 | 8 | 8 | 8 | 8 | 8 | 12 | 10 | 1 | 5 | 0
Not Completed | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Period: Part B- Period 1 (3 Days)
Arm/Group | Placebo: 18-60 Years (HC-HC Diet) | PF-07258669 2 mg: 18-60 Years (HC-HC Diet) | PF-07258669 3 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (HC-HC Diet) | Placebo: 18-60 Years (Standard Diet) | PF-07258669 6 mg: 18-60 Years (Standard Diet) | PF-07258669 20 mg: 18-60 Years (Standard Diet) | PF-07258669 60 mg: 18-60 Years (Standard Diet) | PF-07258669 125 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (Standard Diet) | Placebo: 18-60 Years (HF-HC Diet) | PF-07258669 180 mg: 18-60 Years (HF-HC Diet) | Placebo: Japanese 18-60 Years (Standard Diet) | PF-07258669 180 mg: Japanese 18-60 Years (Standard Diet) | Midazolam Then PF-07258669 + Midazolam: Standard Diet
Started | 0 (No participants for Part B.) | 0 (No participants for Part B.) | 0 (No participants for Part B.) | 0 (No participants for Part B.) | 0 (No participants for Part B.) | 0 (No participants for Part B.) | 0 (No participants for Part B.) | 0 (No participants for Part B.) | 0 (No participants for Part B.) | 0 (No participants for Part B.) | 0 (No participants for Part B.) | 0 (No participants for Part B.) | 0 (No participants for Part B.) | 0 (No participants for Part B.) | 11 (Participants enrolled in Part B of the study.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B- Period 2 (8 Days)
Arm/Group | Placebo: 18-60 Years (HC-HC Diet) | PF-07258669 2 mg: 18-60 Years (HC-HC Diet) | PF-07258669 3 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (HC-HC Diet) | Placebo: 18-60 Years (Standard Diet) | PF-07258669 6 mg: 18-60 Years (Standard Diet) | PF-07258669 20 mg: 18-60 Years (Standard Diet) | PF-07258669 60 mg: 18-60 Years (Standard Diet) | PF-07258669 125 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (Standard Diet) | Placebo: 18-60 Years (HF-HC Diet) | PF-07258669 180 mg: 18-60 Years (HF-HC Diet) | Placebo: Japanese 18-60 Years (Standard Diet) | PF-07258669 180 mg: Japanese 18-60 Years (Standard Diet) | Midazolam Then PF-07258669 + Midazolam: Standard Diet
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who were randomly assigned to study intervention and who took at least 1 dose of study intervention, for the given part of the study (Part A or B).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo: 18-60 Years (HC-HC Diet) | PF-07258669 2 mg: 18-60 Years (HC-HC Diet) | PF-07258669 3 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (HC-HC Diet) | Placebo: 18-60 Years (Standard Diet) | PF-07258669 6 mg: 18-60 Years (Standard Diet) | PF-07258669 20 mg: 18-60 Years (Standard Diet) | PF-07258669 60 mg: 18-60 Years (Standard Diet) | PF-07258669 125 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (Standard Diet) | Placebo: 18-60 Years (HF-HC Diet) | PF-07258669 180 mg: 18-60 Years (HF-HC Diet) | Placebo: Japanese 18-60 Years (Standard Diet) | PF-07258669 180 mg: Japanese 18-60 Years (Standard Diet) | Midazolam Then PF-07258669 + Midazolam: Standard Diet | Total
Number analyzed (Participants) | 6 | 8 | 8 | 7 | 10 | 8 | 8 | 8 | 8 | 8 | 12 | 12 | 1 | 5 | 11 | 120
Age, Customized [Count of Participants; unit: Participants] — Data cannot be reported in 'Placebo: Japanese 18-60 Years (Standard Diet)' reporting group due to risk of re-identification of the participant.
  Participants
    18-44 Years | 2 | 7 | 7 | 6 | 7 | 6 | 5 | 5 | 6 | 7 | 10 | 10 | 0 | 5 | 9 | 92
    45-64 Years | 4 | 1 | 1 | 1 | 3 | 2 | 3 | 3 | 2 | 1 | 2 | 2 | 0 | 0 | 2 | 27
    Not disclosed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Sex/Gender, Customized [Count of Participants; unit: Participants] — Data cannot be reported in 'Placebo: Japanese 18-60 Years (Standard Diet)' reporting group due to risk of re-identification of the participant.
  Participants
    Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Male | 6 | 8 | 8 | 7 | 10 | 8 | 8 | 8 | 7 | 8 | 12 | 12 | 0 | 5 | 11 | 118
    Not disclosed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Data cannot be reported in 'Placebo: Japanese 18-60 Years (Standard Diet)' reporting group due to risk of re-identification of the participant.
  Participants
    Hispanic or Latino | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 8
    Not Hispanic or Latino | 6 | 7 | 7 | 6 | 10 | 8 | 8 | 7 | 5 | 8 | 11 | 12 | 0 | 5 | 10 | 110
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Data cannot be reported in 'Placebo: Japanese 18-60 Years (Standard Diet)' reporting group due to risk of re-identification of the participant.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 5 | 0 | 10
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 1 | 0 | 1 | 3 | 0 | 1 | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 1 | 12
    White | 6 | 6 | 8 | 6 | 7 | 8 | 6 | 8 | 7 | 7 | 7 | 11 | 0 | 0 | 10 | 97
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were events between first dose of study intervention and up to 35 days after last dose of study intervention that were absent before treatment or that worsened after treatment.
Time Frame: Part A: Day 1 to maximum up to 35 days after administration of the final dose of study intervention (maximum up to 49 days)
Population: The safety analysis set for Part A included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention in Part A.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: 18-60 Years (HC-HC Diet) | PF-07258669 2 mg: 18-60 Years (HC-HC Diet) | PF-07258669 3 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (HC-HC Diet) | Placebo: 18-60 Years (Standard Diet) | PF-07258669 6 mg: 18-60 Years (Standard Diet) | PF-07258669 20 mg: 18-60 Years (Standard Diet) | PF-07258669 60 mg: 18-60 Years (Standard Diet) | PF-07258669 125 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (Standard Diet) | Placebo: 18-60 Years (HF-HC Diet) | PF-07258669 180 mg: 18-60 Years (HF-HC Diet) | Placebo: Japanese 18-60 Years (Standard Diet) | PF-07258669 180 mg: Japanese 18-60 Years (Standard Diet)
Number analyzed (Participants) | 6 | 8 | 8 | 7 | 10 | 8 | 8 | 8 | 8 | 8 | 12 | 12 | 1 | 5
Participants | 5 | 8 | 6 | 6 | 9 | 6 | 7 | 4 | 7 | 8 | 8 | 10 | 0 | 3

2. Primary Outcome: Part A: Number of Participants With Laboratory Test Abnormalities Without Regard to Baseline Abnormality
Description: Laboratory assessments included clinical chemistry, hematology, and urinalysis. Abnormality was determined based on the criteria specified in the sponsor reporting standards. The primary criteria was less than (<) 0.8* lower limit of normal (LLN) for lymphocytes and lymphocytes/leukocytes, greater than (>) 1.2* upper limit of normal (ULN) for lymphocytes, eosinophils/leukocytes, monocytes, and monocytes/leukocytes; greater than (>) 3.0* ULN for alanine aminotransferase, >1.3* ULN for urea nitrogen, cholesterol, and triglycerides; >1.030 for specific gravity (scalar), greater than or equal to (>=) 1 for ketones, urine protein, urine hemoglobin, urine bilirubin, leukocyte esterase.
Time Frame: Part A: Baseline to maximum up to 10 days after administration of the final dose of study intervention (maximum up to 24 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: 18-60 Years (HC-HC Diet) | PF-07258669 2 mg: 18-60 Years (HC-HC Diet) | PF-07258669 3 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (HC-HC Diet) | Placebo: 18-60 Years (Standard Diet) | PF-07258669 6 mg: 18-60 Years (Standard Diet) | PF-07258669 20 mg: 18-60 Years (Standard Diet) | PF-07258669 60 mg: 18-60 Years (Standard Diet) | PF-07258669 125 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (Standard Diet) | Placebo: 18-60 Years (HF-HC Diet) | PF-07258669 180 mg: 18-60 Years (HF-HC Diet) | Placebo: Japanese 18-60 Years (Standard Diet) | PF-07258669 180 mg: Japanese 18-60 Years (Standard Diet)
Number analyzed (Participants) | 6 | 8 | 8 | 7 | 10 | 8 | 8 | 8 | 8 | 8 | 12 | 12 | 1 | 5
Participants | 5 | 6 | 6 | 6 | 9 | 5 | 8 | 7 | 8 | 4 | 11 | 8 | 1 | 3

3. Primary Outcome: Part A: Number of Participants With Categorical Summary of Post-Baseline Vital Signs Data
Description: Vital signs included: a) supine systolic blood pressure (SBP): change greater than or equal to (>=) 30 millimeters of mercury (mmHg) increase, postural difference (supine standing) >= 20 mmHg, standing systolic SBP (mmHg) less than (<) 90 mmHg, >= 160 mmHg, change >= 30 mmHg increase, change >= 30 mmHg decrease; b) supine diastolic blood pressure (DBP) < 50 mmHg, >= 90 mmHg, change >= 20 mmHg increase, change >= 20mmHg decrease; postural difference (supine standing) >= 10 mmHg; standing <50 mmHg, value >=90 mmHg, change >=20 mmHg increase, change >=20 mmHg decrease, C) standing pulse rate (PR) greater than (>) 140 bpm. Baseline for supine BP and pulse rate was defined as the average of the triplicate measurements collected at the pre-dose (0 hour) assessment on Day 1. Baseline for standing BP, standing pulse rate, respiratory rate and oral body temperature were defined as the pre-dose (0 hour) assessment on Day 1.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: 18-60 Years (HC-HC Diet) | PF-07258669 2 mg: 18-60 Years (HC-HC Diet) | PF-07258669 3 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (HC-HC Diet) | Placebo: 18-60 Years (Standard Diet) | PF-07258669 6 mg: 18-60 Years (Standard Diet) | PF-07258669 20 mg: 18-60 Years (Standard Diet) | PF-07258669 60 mg: 18-60 Years (Standard Diet) | PF-07258669 125 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (Standard Diet) | Placebo: 18-60 Years (HF-HC Diet) | PF-07258669 180 mg: 18-60 Years (HF-HC Diet) | Placebo: Japanese 18-60 Years (Standard Diet) | PF-07258669 180 mg: Japanese 18-60 Years (Standard Diet)
Number analyzed (Participants) | 6 | 8 | 8 | 7 | 10 | 8 | 8 | 8 | 8 | 8 | 12 | 12 | 1 | 5
Participants
  Supine SBP Change >= 30mmHg increase | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SBP postural difference >=20mmHg | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Standing SBP Value < 90 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
  Standing SBP Value >= 160 mmHg | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 0
  Standing SBP Value >= 30 mmHg increase | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 3 | 3 | 0 | 1
  Standing SBP Value >= 30 mmHg decrease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Supine DBP Value >= 30 mmHg decrease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Supine DBP value < 50 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Supine DBP value >= 90 mmHg | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine DBP change >= 20 mmHg increase | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine DBP change >= 20 mmHg decrease | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DBP (mmHg) postural difference (supine standing) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0
  Standing DBP value < 50 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Standing DBP value >= 90 mmHg | 2 | 4 | 1 | 1 | 3 | 1 | 3 | 3 | 1 | 0 | 3 | 2 | 0 | 0
  Standing DBP change >= 20 mmHg increase | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 0
  Standing diastolic BP change >= 20 mmHg decrease | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 0
  Standing PR >140 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Part A: Number of Participants Who Met Defined Electrocardiogram (ECG) Criteria
Description: ECG criteria: QTc corrected using Fridericia's formula (QTCF) interval aggregate in milliseconds (msec): less than or equal to (<=) change <= 60 msec. Baseline was defined as the average of the triplicate ECG measurements over the 3 pre-dose measurement times (-1 hour, -0.5 hour, and pre-dose 0 hour; total of 9 ECG measurements) on Day 1.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: 18-60 Years (HC-HC Diet) | PF-07258669 2 mg: 18-60 Years (HC-HC Diet) | PF-07258669 3 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (HC-HC Diet) | Placebo: 18-60 Years (Standard Diet) | PF-07258669 6 mg: 18-60 Years (Standard Diet) | PF-07258669 20 mg: 18-60 Years (Standard Diet) | PF-07258669 60 mg: 18-60 Years (Standard Diet) | PF-07258669 125 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (Standard Diet) | Placebo: 18-60 Years (HF-HC Diet) | PF-07258669 180 mg: 18-60 Years (HF-HC Diet) | Placebo: Japanese 18-60 Years (Standard Diet) | PF-07258669 180 mg: Japanese 18-60 Years (Standard Diet)
Number analyzed (Participants) | 6 | 8 | 8 | 7 | 10 | 8 | 8 | 8 | 8 | 8 | 12 | 12 | 1 | 5
Participants | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0

5. Primary Outcome: Part A: Number of Participants With Positive Response on Columbia Suicide Severity Rating Scale (C-SSRS) at Screening
Description: C-SSRS is interview-based rating scale to assess suicidal ideation and behavior. C-SSRS was mapped to Columbia-Classification Algorithm of Suicide Assessment(C-CASA) and suicidal behavior events were scored as follows:1.Completed suicide,2.Suicide attempt,3.Interrupted attempt,4.Aborted attempt,5.Preparatory actions toward imminent suicidal behaviors. Participants with response "Yes" to items 4,5 or behavioral question of C-SSRS were assessed by clinician and had their suicidality managed. Suicidal behaviors were scored as1.Completed suicide response "Yes" on "Completed Suicide",2.Suicide attempt had response "Yes" on "Actual Attempt",3.Interrupted attempt, had response "Yes" on "Interrupted attempt",4.Aborted attempt, had response "Yes" on "Aborted attempt",5.Preparatory actions toward imminent suicidal behaviors, had response "Yes" on "Preparatory Acts or Behavior".Here, number of participants with positive response (response of "yes") to suicidal behavior or ideation were reported.
Time Frame: Part A: At Screening (Day-28 [28 days prior to dosing] to Day -3 [3 days prior to dosing])
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: 18-60 Years (HC-HC Diet) | PF-07258669 2 mg: 18-60 Years (HC-HC Diet) | PF-07258669 3 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (HC-HC Diet) | Placebo: 18-60 Years (Standard Diet) | PF-07258669 6 mg: 18-60 Years (Standard Diet) | PF-07258669 20 mg: 18-60 Years (Standard Diet) | PF-07258669 60 mg: 18-60 Years (Standard Diet) | PF-07258669 125 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (Standard Diet) | Placebo: 18-60 Years (HF-HC Diet) | PF-07258669 180 mg: 18-60 Years (HF-HC Diet) | Placebo: Japanese 18-60 Years (Standard Diet) | PF-07258669 180 mg: Japanese 18-60 Years (Standard Diet)
Number analyzed (Participants) | 6 | 8 | 8 | 7 | 10 | 8 | 8 | 8 | 8 | 8 | 12 | 12 | 1 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Part A: Number of Participants With Positive Response on Columbia Suicide Severity Rating Scale (C-SSRS) on Day -2
Description: as for outcome 5
Time Frame: Part A: On Day -2 (2 days prior to dosing)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: 18-60 Years (HC-HC Diet) | PF-07258669 2 mg: 18-60 Years (HC-HC Diet) | PF-07258669 3 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (HC-HC Diet) | Placebo: 18-60 Years (Standard Diet) | PF-07258669 6 mg: 18-60 Years (Standard Diet) | PF-07258669 20 mg: 18-60 Years (Standard Diet) | PF-07258669 60 mg: 18-60 Years (Standard Diet) | PF-07258669 125 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (Standard Diet) | Placebo: 18-60 Years (HF-HC Diet) | PF-07258669 180 mg: 18-60 Years (HF-HC Diet) | Placebo: Japanese 18-60 Years (Standard Diet) | PF-07258669 180 mg: Japanese 18-60 Years (Standard Diet)
Number analyzed (Participants) | 6 | 8 | 8 | 7 | 10 | 8 | 8 | 8 | 8 | 8 | 12 | 12 | 1 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Part A: Number of Participants With Positive Response on Columbia Suicide Severity Rating Scale (C-SSRS) on Day 7
Description: as for outcome 5
Time Frame: Part A: On Day 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: 18-60 Years (HC-HC Diet) | PF-07258669 2 mg: 18-60 Years (HC-HC Diet) | PF-07258669 3 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (HC-HC Diet) | Placebo: 18-60 Years (Standard Diet) | PF-07258669 6 mg: 18-60 Years (Standard Diet) | PF-07258669 20 mg: 18-60 Years (Standard Diet) | PF-07258669 60 mg: 18-60 Years (Standard Diet) | PF-07258669 125 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (Standard Diet) | Placebo: 18-60 Years (HF-HC Diet) | PF-07258669 180 mg: 18-60 Years (HF-HC Diet) | Placebo: Japanese 18-60 Years (Standard Diet) | PF-07258669 180 mg: Japanese 18-60 Years (Standard Diet)
Number analyzed (Participants) | 6 | 8 | 8 | 7 | 10 | 8 | 8 | 8 | 8 | 8 | 12 | 12 | 1 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Part A: Number of Participants With Positive Response on Columbia Suicide Severity Rating Scale (C-SSRS) on Day 14
Description: as for outcome 5
Time Frame: Part A: Day 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: 18-60 Years (HC-HC Diet) | PF-07258669 2 mg: 18-60 Years (HC-HC Diet) | PF-07258669 3 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (HC-HC Diet) | Placebo: 18-60 Years (Standard Diet) | PF-07258669 6 mg: 18-60 Years (Standard Diet) | PF-07258669 20 mg: 18-60 Years (Standard Diet) | PF-07258669 60 mg: 18-60 Years (Standard Diet) | PF-07258669 125 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (Standard Diet) | Placebo: 18-60 Years (HF-HC Diet) | PF-07258669 180 mg: 18-60 Years (HF-HC Diet) | Placebo: Japanese 18-60 Years (Standard Diet) | PF-07258669 180 mg: Japanese 18-60 Years (Standard Diet)
Number analyzed (Participants) | 6 | 8 | 8 | 7 | 10 | 8 | 8 | 8 | 8 | 8 | 12 | 12 | 1 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Part A: Number of Participants With Positive Response on Columbia Suicide Severity Rating Scale (C-SSRS) on Day 21
Description: as for outcome 5
Time Frame: Part A: Day 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: 18-60 Years (HC-HC Diet) | PF-07258669 2 mg: 18-60 Years (HC-HC Diet) | PF-07258669 3 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (HC-HC Diet) | Placebo: 18-60 Years (Standard Diet) | PF-07258669 6 mg: 18-60 Years (Standard Diet) | PF-07258669 20 mg: 18-60 Years (Standard Diet) | PF-07258669 60 mg: 18-60 Years (Standard Diet) | PF-07258669 125 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (Standard Diet) | Placebo: 18-60 Years (HF-HC Diet) | PF-07258669 180 mg: 18-60 Years (HF-HC Diet) | Placebo: Japanese 18-60 Years (Standard Diet) | PF-07258669 180 mg: Japanese 18-60 Years (Standard Diet)
Number analyzed (Participants) | 6 | 8 | 8 | 7 | 10 | 8 | 8 | 8 | 8 | 8 | 12 | 12 | 1 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Part A: Number of Participants With 24-Hour Fluid Intake and Urine Output >6 Liters Per Day at Screening
Description: All fluids consumed by the participants between 0 to 24 hours on days requiring 24-hour fluid intake assessments were recorded by clinical research unit (CRU) staff. The cumulative fluid intake for the 24-hour period was measured and recorded. Participants were instructed to void urine to empty their bladder at 0 hours. All urine voided after this time was collected up to, and including, a final void of urine at 24 hours.
Time Frame: Part A: At Screening (Day-28 [28 days prior to dosing] to Day -3 [3 days prior to dosing])
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: 18-60 Years (HC-HC Diet) | PF-07258669 2 mg: 18-60 Years (HC-HC Diet) | PF-07258669 3 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (HC-HC Diet) | Placebo: 18-60 Years (Standard Diet) | PF-07258669 6 mg: 18-60 Years (Standard Diet) | PF-07258669 20 mg: 18-60 Years (Standard Diet) | PF-07258669 60 mg: 18-60 Years (Standard Diet) | PF-07258669 125 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (Standard Diet) | Placebo: 18-60 Years (HF-HC Diet) | PF-07258669 180 mg: 18-60 Years (HF-HC Diet) | Placebo: Japanese 18-60 Years (Standard Diet) | PF-07258669 180 mg: Japanese 18-60 Years (Standard Diet)
Number analyzed (Participants) | 6 | 8 | 8 | 7 | 10 | 8 | 8 | 8 | 8 | 8 | 12 | 12 | 1 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Primary Outcome: Part A: Number of Participants With 24-Hour Fluid Intake and Urine Output >6 Liters Per Day on Day -1
Description: All fluids consumed by the participants between 0 to 24 hours on days requiring 24-hour fluid intake assessments were recorded by CRU staff. The cumulative fluid intake for the 24-hour period was measured and recorded. Participants were instructed to void urine to empty their bladder at 0 hours. All urine voided after this time was collected up to, and including, a final void of urine at 24 hours.
Time Frame: Part A: Day -1 (1 day prior to dosing)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: 18-60 Years (HC-HC Diet) | PF-07258669 2 mg: 18-60 Years (HC-HC Diet) | PF-07258669 3 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (HC-HC Diet) | Placebo: 18-60 Years (Standard Diet) | PF-07258669 6 mg: 18-60 Years (Standard Diet) | PF-07258669 20 mg: 18-60 Years (Standard Diet) | PF-07258669 60 mg: 18-60 Years (Standard Diet) | PF-07258669 125 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (Standard Diet) | Placebo: 18-60 Years (HF-HC Diet) | PF-07258669 180 mg: 18-60 Years (HF-HC Diet) | Placebo: Japanese 18-60 Years (Standard Diet) | PF-07258669 180 mg: Japanese 18-60 Years (Standard Diet)
Number analyzed (Participants) | 6 | 8 | 8 | 7 | 10 | 8 | 8 | 8 | 8 | 8 | 12 | 12 | 1 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: Part A: Number of Participants With 24-Hour Fluid Intake and Urine Output >6 Liters Per Day on Day 7
Description: as for outcome 11
Time Frame: Part A: Day 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: 18-60 Years (HC-HC Diet) | PF-07258669 2 mg: 18-60 Years (HC-HC Diet) | PF-07258669 3 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (HC-HC Diet) | Placebo: 18-60 Years (Standard Diet) | PF-07258669 6 mg: 18-60 Years (Standard Diet) | PF-07258669 20 mg: 18-60 Years (Standard Diet) | PF-07258669 60 mg: 18-60 Years (Standard Diet) | PF-07258669 125 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (Standard Diet) | Placebo: 18-60 Years (HF-HC Diet) | PF-07258669 180 mg: 18-60 Years (HF-HC Diet) | Placebo: Japanese 18-60 Years (Standard Diet) | PF-07258669 180 mg: Japanese 18-60 Years (Standard Diet)
Number analyzed (Participants) | 6 | 8 | 8 | 7 | 10 | 8 | 8 | 8 | 8 | 8 | 12 | 12 | 1 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Primary Outcome: Part A: Number of Participants With 24-Hour Fluid Intake and Urine Output >6 Liters Per Day on Day 14
Description: as for outcome 11
Time Frame: Part A: Day 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: 18-60 Years (HC-HC Diet) | PF-07258669 2 mg: 18-60 Years (HC-HC Diet) | PF-07258669 3 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (HC-HC Diet) | Placebo: 18-60 Years (Standard Diet) | PF-07258669 6 mg: 18-60 Years (Standard Diet) | PF-07258669 20 mg: 18-60 Years (Standard Diet) | PF-07258669 60 mg: 18-60 Years (Standard Diet) | PF-07258669 125 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (Standard Diet) | Placebo: 18-60 Years (HF-HC Diet) | PF-07258669 180 mg: 18-60 Years (HF-HC Diet) | Placebo: Japanese 18-60 Years (Standard Diet) | PF-07258669 180 mg: Japanese 18-60 Years (Standard Diet)
Number analyzed (Participants) | 6 | 8 | 8 | 7 | 10 | 8 | 8 | 8 | 8 | 8 | 12 | 12 | 1 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Primary Outcome: Part B: Maximum Observed Plasma Concentration (Cmax) of Midazolam Alone on Day 1 of Period 1
Description: Cmax was defined as the maximum observed plasma concentration.
Time Frame: Part B/Period 1: 0.5, 1, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Day 1
Population: Pharmacokinetic (PK) parameter set included all participants randomly assigned to study intervention and who took at least 1 dose of midazolam and had at least one of the PK parameters of interest calculated, for Part B of the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Groups:
- Part B Period 1: Midazolam: Healthy non-Japanese participants aged 18-60 years who were on standard diet, received midazolam 1 mg oral solution on Day 1 of Period 1.
Arm/Group | Part B Period 1: Midazolam
Number analyzed (Participants) | 11
Nanogram per milliliter | 6.213 (43)

15. Primary Outcome: Part B: Cmax of Midazolam in Combination With PF-07258669 on Day 2 of Period 2
Description: Cmax is the maximum observed plasma concentration.
Time Frame: Part B/Period 2: 0.5, 1, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Day 2
Population: PK parameter set included all participants randomly assigned to study intervention and who took at least 1 dose of midazolam and had at least one of the PK parameters of interest calculated, for Part B of the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Groups:
- Part B Period 2: PF-07258669 + Midazolam (Day 2): Healthy non-Japanese participants aged 18-60 years who were on standard diet, received oral PF-07258669 180 mg tablets, Q8H from Day 1 to Day 10 of Period 2. On Days 2 and 10 of Period 2, participants received midazolam 1 mg oral solution.
Arm/Group | Part B Period 2: PF-07258669 + Midazolam (Day 2)
Number analyzed (Participants) | 11
Nanogram per milliliter | 10.83 (27)

16. Primary Outcome: Part B: Cmax of Midazolam in Combination With PF-07258669 on Day 10 of Period 2
Description: Cmax was defined as the maximum observed plasma concentration.
Time Frame: Part B/Period 2: 0.5, 1, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Day 10
Population: PK parameter set included all participants randomly assigned to study intervention and who took at least 1 dose of midazolam and had at least one of the PK parameters of interest calculated, for Part B of the study. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Groups:
- Part B Period 2: PF-07258669 + Midazolam (Day 10): Healthy non-Japanese participants aged 18-60 years who were on standard diet, received oral PF-07258669 180 mg tablets, Q8H from Day 1 to Day 10 of Period 2. On Day 10 of Period 2, participants received midazolam 1 mg oral solution.
Arm/Group | Part B Period 2: PF-07258669 + Midazolam (Day 10)
Number analyzed (Participants) | 9
Nanogram per milliliter | 11.73 (30)

17. Primary Outcome: Part B: Area Under the Plasma Concentration-Time Curve From Time Zero (0) to the Time of the Last Quantifiable Concentration (AUClast) of Midazolam Alone on Day 1 of Period 1
Description: AUClast was the area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration.
Time Frame: Part B/Period 1: 0.5, 1, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Day 1
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Part B Period 1: Midazolam
Number analyzed (Participants) | 11
Nanogram*hour per milliliter | 18.56 (47)

18. Primary Outcome: Part B: AUClast of Midazolam in Combination With PF-07258669 on Day 2 of Period 2
Description: AUClast was defined as the area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration.
Time Frame: Part B/Period 2: 0.5, 1, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Day 2
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Groups:
- Part B Period 2: PF-07258669 + Midazolam (Day 2): Healthy non-Japanese participants aged 18-60 years who were on standard diet, received oral PF-07258669 180 mg tablets, Q8H from Day 1 to Day 10 of Period 2. On Day 2 of Period 2, participants received midazolam 1 mg oral solution.
Arm/Group | Part B Period 2: PF-07258669 + Midazolam (Day 2)
Number analyzed (Participants) | 11
Nanogram*hour per milliliter | 30.27 (35)

19. Primary Outcome: Part B: AUClast of Midazolam in Combination With PF-07258669 on Day 10 of Period 2
Description: as for outcome 18
Time Frame: Part B/ Period 2: 0.5, 1, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Day 10
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Part B Period 2: PF-07258669 + Midazolam (Day 10)
Number analyzed (Participants) | 9
Nanogram*hour per milliliter | 40.41 (33)

20. Primary Outcome: Part B: Area Under the Plasma Concentration-Time Curve From Time 0 to Extrapolated Infinite Time (AUCinf) of Midazolam Alone on Day 1 of Period 1
Description: AUCinf was defined as the area under the plasma concentration time profile from time 0 extrapolated to infinite time.
Time Frame: Part B/Period 1: 0.5, 1, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Day 1
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Part B Period 1: Midazolam
Number analyzed (Participants) | 10
Nanogram*hour per milliliter | 19.35 (48)

21. Primary Outcome: Part B: AUCinf of Midazolam in Combination With PF-07258669 on Day 2 of Period 2
Description: AUCinf was defined as the area under the plasma concentration time profile from time 0 extrapolated to infinite time.
Time Frame: Part B/Period 2: 0.5, 1, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Day 2
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Part B Period 2: PF-07258669 + Midazolam (Day 2)
Number analyzed (Participants) | 10
Nanogram*hour per milliliter | 32.84 (32)

22. Primary Outcome: Part B: AUCinf of Midazolam in Combination With PF-07258669 on Day 10 of Period 2
Description: AUCinf was defined as the area under the plasma concentration time profile from time 0 extrapolated to infinite time.
Time Frame: Part B/ Period 2: 0.5, 1, 2, 3, 4, 6, 8, 10, 12, and 16 hours post-dose on Day 10
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Part B Period 2: PF-07258669 + Midazolam (Day 10)
Number analyzed (Participants) | 9
Nanogram*hour per milliliter | 41.16 (34)

23. Secondary Outcome: Part A: Maximum Observed Plasma Concentration (Cmax) of PF-07258669 on Days 1 and 14
Description: Cmax was defined as the maximum plasma concentration.
Time Frame: Part A: 0, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 hours post dose on Day 1 and Day 14
Population: PK parameter set included all participants randomly assigned to study intervention and who took at least 1 dose of midazolam and/or study intervention and had at least one of the PK parameters of interest calculated, for part A of the study. Here, 'Number Analyzed' signifies participants evaluable for the specified rows.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | PF-07258669 2 mg: 18-60 Years (HC-HC Diet) | PF-07258669 3 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (Standard Diet) | PF-07258669 20 mg: 18-60 Years (Standard Diet) | PF-07258669 60 mg: 18-60 Years (Standard Diet) | PF-07258669 125 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (HF-HC Diet) | PF-07258669 180 mg: Japanese 18-60 Years (Standard Diet)
Number analyzed (Participants) | 8 | 8 | 7 | 8 | 8 | 8 | 8 | 8 | 12 | 5
Nanogram per milliliter
  Day 1 | 19.47 (25) | 25.06 (22) | 50.41 (22) | 45.99 (47) | 131.2 (32) | 468.3 (27) | 987.2 (28) | 1263 (37) | 1218 (42) | 1210 (9)
  Day 14: number analyzed (Participants) | 8 | 8 | 6 | 8 | 8 | 8 | 8 | 8 | 10 | 5
  Day 14 | 21.96 (21) | 27.91 (25) | 59.76 (29) | 57.08 (39) | 165.2 (25) | 568.5 (26) | 1246 (25) | 1464 (21) | 1772 (19) | 1750 (26)

24. Secondary Outcome: Part A: Dose Normalized Maximum Observed Plasma Concentration (Cmax,dn) of PF-07258669 on Days 1 and 14
Description: Cmax was defined maximum observed serum concentration. Cmax (dn) was calculated as Cmax/dose.
Time Frame: Part A: 0, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 hours post dose on Day 1 and Day 14
Population: PK analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of midazolam and/or study intervention and had at least one of the PK parameters of interest calculated, for part A of the study. Here, 'Number Analyzed' signifies participants evaluable for the specified rows.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter per milligram
Arm/Group | PF-07258669 2 mg: 18-60 Years (HC-HC Diet) | PF-07258669 3 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (Standard Diet) | PF-07258669 20 mg: 18-60 Years (Standard Diet) | PF-07258669 60 mg: 18-60 Years (Standard Diet) | PF-07258669 125 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (HF-HC Diet) | PF-07258669 180 mg: Japanese 18-60 Years (Standard Diet)
Number analyzed (Participants) | 8 | 8 | 7 | 8 | 8 | 8 | 8 | 8 | 12 | 5
Nanograms per milliliter per milligram
  Day 1 | 9.742 (25) | 8.352 (22) | 8.403 (22) | 7.666 (47) | 6.562 (32) | 7.803 (27) | 7.899 (28) | 7.013 (37) | 6.770 (42) | 6.719 (9)
  Day 14: number analyzed (Participants) | 8 | 7 | 6 | 8 | 8 | 8 | 8 | 8 | 12 | 5
  Day 14 | 10.99 (22) | 9.301 (25) | 9.952 (29) | 9.515 (39) | 8.269 (25) | 9.473 (26) | 9.982 (25) | 8.134 (22) | 9.849 (19) | 9.723 (26)

25. Secondary Outcome: Part A: Area Under the Plasma Concentration-Time Curve From Time 0 to Dosing Interval (Tau) (AUCtau) of PF-07258669 on Days 1 and 14
Description: Area under the plasma concentration-time profile from time zero to time tau, the dosing interval, where tau = 8 hours.
Time Frame: Part A: 0 to 8, 8 to 16, and 16 to 24 hours post dose on Day 1 and Day 14
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms*hours per (/) milliliter
Arm/Group | PF-07258669 2 mg: 18-60 Years (HC-HC Diet) | PF-07258669 3 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (Standard Diet) | PF-07258669 20 mg: 18-60 Years (Standard Diet) | PF-07258669 60 mg: 18-60 Years (Standard Diet) | PF-07258669 125 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (HF-HC Diet) | PF-07258669 180 mg: Japanese 18-60 Years (Standard Diet)
Number analyzed (Participants) | 8 | 8 | 7 | 8 | 8 | 8 | 8 | 8 | 12 | 5
Nanograms*hours per (/) milliliter
  Day 1 | 46.27 (26) | 60.42 (27) | 113.6 (15) | 107.2 (42) | 388.1 (38) | 1207 (26) | 2597 (29) | 3357 (34) | 3361 (27) | 3331 (13)
  Day 14: number analyzed (Participants) | 8 | 7 | 6 | 8 | 8 | 8 | 8 | 8 | 10 | 5
  Day 14 | 62.40 (32) | 76.25 (30) | 162.0 (28) | 147.0 (45) | 480.4 (28) | 1795 (26) | 3946 (28) | 5313 (31) | 5845 (19) | 6074 (21)

26. Secondary Outcome: Part A: Dose Normalized Area Under the Curve From Time 0 to Dosing Interval (Tau) (AUCtau, dn) of PF-07258669 on Days 1 and 14
Time Frame: Part A: 0 to 8, 8 to 16, and 16 to 24 hours post dose on Day 1 and Day 14
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms*hours/ milliliter/ milligrams
Arm/Group | PF-07258669 2 mg: 18-60 Years (HC-HC Diet) | PF-07258669 3 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (Standard Diet) | PF-07258669 20 mg: 18-60 Years (Standard Diet) | PF-07258669 60 mg: 18-60 Years (Standard Diet) | PF-07258669 125 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (HF-HC Diet) | PF-07258669 180 mg: Japanese 18-60 Years (Standard Diet)
Number analyzed (Participants) | 8 | 8 | 7 | 8 | 8 | 8 | 8 | 8 | 12 | 5
Nanograms*hours/ milliliter/ milligrams
  Day 1 | 23.16 (26) | 20.15 (27) | 18.93 (15) | 17.87 (42) | 19.42 (38) | 20.14 (26) | 20.75 (29) | 18.64 (34) | 18.67 (27) | 18.52 (13)
  Day 14: number analyzed (Participants) | 8 | 7 | 6 | 8 | 8 | 8 | 8 | 8 | 10 | 5
  Day 14 | 31.21 (32) | 25.44 (30) | 27.01 (28) | 24.47 (45) | 24.04 (28) | 29.90 (26) | 31.57 (28) | 29.49 (31) | 32.49 (19) | 33.74 (21)

27. Secondary Outcome: Part A: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-07258669 on Days 1 and 14
Description: Tmax was defined as the time taken (in hours) to reach the maximum plasma drug concentration.
Time Frame: Part A: 0, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 hours post dose on Day 1 and Day 14
Population: as for outcome 24
Measure: Median (Full Range); unit: Hours
Arm/Group | PF-07258669 2 mg: 18-60 Years (HC-HC Diet) | PF-07258669 3 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (Standard Diet) | PF-07258669 20 mg: 18-60 Years (Standard Diet) | PF-07258669 60 mg: 18-60 Years (Standard Diet) | PF-07258669 125 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (HF-HC Diet) | PF-07258669 180 mg: Japanese 18-60 Years (Standard Diet)
Number analyzed (Participants) | 8 | 8 | 7 | 8 | 8 | 8 | 8 | 8 | 12 | 5
Hours
  Day 1 | 1.000 [0.500 to 1.50] | 1.000 [0.500 to 1.05] | 0.5830 [0.500 to 1.50] | 0.8265 [0.500 to 1.13] | 1.010 [0.500 to 2.00] | 1.000 [0.500 to 1.50] | 1.000 [0.500 to 1.50] | 1.000 [1.00 to 1.05] | 1.000 [0.550 to 1.50] | 0.5830 [0.500 to 1.50]
  Day 14: number analyzed (Participants) | 8 | 7 | 6 | 8 | 8 | 8 | 8 | 8 | 10 | 5
  Day 14 | 1.010 [0.500 to 1.52] | 1.000 [0.500 to 1.02] | 0.7415 [0.500 to 1.50] | 0.7665 [0.500 to 1.07] | 1.000 [1.00 to 1.53] | 1.000 [0.500 to 1.05] | 1.000 [0.500 to 1.08] | 1.500 [1.00 to 2.00] | 1.000 [0.500 to 1.50] | 1.000 [1.00 to 1.02]

28. Secondary Outcome: Part A: Amount of PF-0728669 Excreted Unchanged in Urine Over the Dosing Interval Tau (Aetau)
Description: Aetau was defined as the amount of unchanged drug recovered in urine during the dosing interval.
Time Frame: Part A: 0 to 8, 8 to 16, and 16 to 24 hours post dose on Day 14
Population: PK analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of midazolam and/or study intervention and had at least one of the PK parameters of interest calculated, for part A of the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligrams
Arm/Group | PF-07258669 2 mg: 18-60 Years (HC-HC Diet) | PF-07258669 3 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (Standard Diet) | PF-07258669 20 mg: 18-60 Years (Standard Diet) | PF-07258669 60 mg: 18-60 Years (Standard Diet) | PF-07258669 125 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (HF-HC Diet) | PF-07258669 180 mg: Japanese 18-60 Years (Standard Diet)
Number analyzed (Participants) | 8 | 8 | 7 | 8 | 8 | 8 | 8 | 8 | 12 | 5
Milligrams | 0.004304 (45) | 0.004490 (153) | 0.01690 (34) | 0.01462 (49) | 0.04039 (70) | 0.1440 (43) | 0.3173 (109) | 0.3371 (188) | 0.3146 (314) | 0.6581 (37)

29. Secondary Outcome: Part A: Percentage Dose of PF-07258669 Excreted Unchanged in the Urine Over the Dosing Interval Tau (Aetau%)
Description: Aetau% was defined as the percentage of dose recovered in urine as unchanged drug.
Time Frame: Part A: 0 to 8, 8 to 16, and 16 to 24 hours post dose on Day 14
Population: as for outcome 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of dose
Arm/Group | PF-07258669 2 mg: 18-60 Years (HC-HC Diet) | PF-07258669 3 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (Standard Diet) | PF-07258669 20 mg: 18-60 Years (Standard Diet) | PF-07258669 60 mg: 18-60 Years (Standard Diet) | PF-07258669 125 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (HF-HC Diet) | PF-07258669 180 mg: Japanese 18-60 Years (Standard Diet)
Number analyzed (Participants) | 8 | 8 | 7 | 8 | 8 | 8 | 8 | 8 | 12 | 5
Percentage of dose | 0.2152 (45) | 0.1496 (153) | 0.2814 (34) | 0.2436 (49) | 0.2020 (70) | 0.2400 (43) | 0.2536 (109) | 0.1872 (189) | 0.1748 (314) | 0.3654 (37)

30. Secondary Outcome: Part A: Renal Clearance (CLr) of PF-07258669
Description: Renal clearance was calculated as cumulative amount of drug recovered unchanged in urine during the dosing interval (Aetau) divided by area under the plasma concentration time-curve from time zero to end of dosing interval (AUCtau).
Time Frame: Part A: 0 to 8, 8 to 16, and 16 to 24 hours post dose on Day 14
Population: as for outcome 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/ hour
Arm/Group | PF-07258669 2 mg: 18-60 Years (HC-HC Diet) | PF-07258669 3 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (Standard Diet) | PF-07258669 20 mg: 18-60 Years (Standard Diet) | PF-07258669 60 mg: 18-60 Years (Standard Diet) | PF-07258669 125 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (HF-HC Diet) | PF-07258669 180 mg: Japanese 18-60 Years (Standard Diet)
Number analyzed (Participants) | 8 | 8 | 7 | 8 | 8 | 8 | 8 | 8 | 12 | 5
Liter/ hour | 0.06896 (37) | 0.05887 (171) | 0.1042 (44) | 0.09946 (33) | 0.08412 (48) | 0.08026 (55) | 0.08040 (116) | 0.06341 (241) | 0.05381 (350) | 0.1083 (31)

31. Secondary Outcome: Part B: Number of Participants With TEAEs
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were events between first dose of study drug and up to follow-up visit that were absent before treatment or that worsened after treatment.
Time Frame: Part B: Day 1 to maximum up to 35 days after administration of the final dose of study intervention (maximum up to 46 days)
Population: The safety analysis set for Part B included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention in Part B.
Measure: Count of Participants; unit: Participants
Groups:
- Part B Period 2: PF-07258669 + Midazolam (Day 2): Healthy non-Japanese participants aged 18-60 years who were on standard diet, received oral PF-07258669 180 mg tablets Q8H from Day 1 to 10 of Period 2. On day 2 of Period 2, participants received midazolam 1 mg oral solution.
- Part B Period 2: PF-07258669 + Midazolam (Day 10): Healthy non-Japanese participants aged 18-60 years who were on standard diet, received oral PF-07258669 180 mg tablets Q8H from Day 1 to 10 of Period 2. On day 10 of Period 2, participants received midazolam 1 mg oral solution.
Arm/Group | Part B Period 1: Midazolam | Part B Period 2: PF-07258669 + Midazolam (Day 2) | Part B Period 2: PF-07258669 + Midazolam (Day 10)
Number analyzed (Participants) | 11 | 11 | 9
Participants | 2 | 8 | 2

32. Secondary Outcome: Part B: Number of Participants With Categorical Summary of Post-Baseline Vital Signs Data
Description: Vital signs examination included: supine systolic blood pressure with criteria change >= 30 mmHg decrease, supine diastolic blood pressure with criteria value >= 90 mmHg and change >= 20 mmHg decrease.
Time Frame: Part B: Day 1 of Period 1 up to Day 10 of Period 2 (12 days)
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Part B Period 1: Midazolam | Part B Period 2: PF-07258669 + Midazolam (Day 2) | Part B Period 2: PF-07258669 + Midazolam (Day 10)
Number analyzed (Participants) | 11 | 11 | 9
Participants
  Standing systolic blood pressure | 0 | 1 | 1
  Standing diastolic blood pressure: value >= 90 mmHg | 0 | 1 | 1
  Standing diastolic blood pressure: value change >= 20 mmHg decrease | 0 | 2 | 1

33. Secondary Outcome: Part B: Number of Participants Who Met Defined Electrocardiogram (ECG) Criteria
Description: Following ECG parameters were analyzed: QTCF interval with criteria 450 less than (<) value less than or equal to (<=) 480. A standard 12-lead ECGs utilizing limb leads were collected using an ECG machine that automatically calculated the heart rate and measures PR, QT, and QTc intervals and QRS complex. On Day 1 at -1 hour (h), -0.5h, and 0h prior to the morning dose, triplicate 12-lead ECGs were obtained approximately 2 to 4 minutes apart at each time point. The average of the triplicate ECG measurements over the 3 pre dose measurement times (total of 9 ECG measurements) collected before morning dose administration on Day 1 served as each participant's baseline QTc value.
Time Frame: Part B: Day 1 of Period 1 up to Day 10 of Period 2 (12 days)
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Part B Period 1: Midazolam | Part B Period 2: PF-07258669 + Midazolam (Day 2) | Part B Period 2: PF-07258669 + Midazolam (Day 10)
Number analyzed (Participants) | 11 | 11 | 9
Participants | 0 | 0 | 1

34. Secondary Outcome: Part B: Number of Participants With Laboratory Test Abnormalities Without Regard to Baseline Abnormality
Description: Laboratory parameters assessed included: hematology (monocytes, monocytes/leukocytes) with primary criteria greater than (>) 1.2*upper limit of normal (ULN), clinical chemistry (bilirubin, direct bilirubin and indirect bilirubin with primary criteria >1.5*ULN, alanine aminotransferase with primary criteria >3.0*ULN, creatine kinase with primary criteria >2.0*ULN, urobilinogen with primary criteria greater than or equal to (>=)1, cholesterol and triglycerides-fasting with primary criteria >1.3*ULN), urinalysis (ketones and urine hemoglobin with primary criteria >=1).
Time Frame: as for outcome 31
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Part B Period 1: Midazolam | Part B Period 2: PF-07258669 + Midazolam (Day 2) | Part B Period 2: PF-07258669 + Midazolam (Day 10)
Number analyzed (Participants) | 11 | 11 | 9
Participants | 2 | 4 | 4

ADVERSE EVENTS:
Time Frame: Part A: Day 1 to maximum up to 35 days after administration of the final dose of study intervention (maximum up to 49 days), Part B: Day 1 to maximum up to 35 days after administration of the final dose of study intervention (maximum up to 46 days)
Description: Safety analysis set included all participants who were randomly assigned to study intervention and who took at least 1 dose of study intervention, for the given part of the study (Part A or B). Participants were analyzed according to the product they received.
Arm/Group | Placebo: 18-60 Years (HC-HC Diet) | PF-07258669 2 mg: 18-60 Years (HC-HC Diet) | PF-07258669 3 mg: 18-60 Years (HC-HC Diet) | PF-07258669 6 mg: 18-60 Years (HC-HC Diet) | Placebo: 18-60 Years (Standard Diet) | PF-07258669 6 mg: 18-60 Years (Standard Diet) | PF-07258669 20 mg: 18-60 Years (Standard Diet) | PF-07258669 60 mg: 18-60 Years (Standard Diet) | PF-07258669 125 mg: 18-60 Years (Standard Diet) | PF-07258669 180 mg: 18-60 Years (Standard Diet) | Placebo: 18-60 Years (HF-HC Diet) | PF-07258669 180 mg: 18-60 Years (HF-HC Diet) | Placebo: Japanese 18-60 Years (Standard Diet) | PF-07258669 180 mg: Japanese 18-60 Years (Standard Diet) | Part B Period 1: Midazolam | Part B Period 2: PF-07258669 + Midazolam (Day 2) | Part B Period 2: PF-07258669 + Midazolam (Day 10)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8 | 0/8 | 0/7 | 0/10 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/12 | 0/12 | 0/1 | 0/5 | 0/11 | 0/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 1/8 | 0/7 | 0/10 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/12 | 0/12 | 0/1 | 0/5 | 0/11 | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 5/6 | 8/8 | 6/8 | 6/7 | 9/10 | 6/8 | 7/8 | 4/8 | 7/8 | 8/8 | 8/12 | 10/12 | 0/1 | 3/5 | 2/11 | 8/11 | 2/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo: 18-60 Years (HC-HC Diet) (N=6) | PF-07258669 2 mg: 18-60 Years (HC-HC Diet) (N=8) | PF-07258669 3 mg: 18-60 Years (HC-HC Diet) (N=8) | PF-07258669 6 mg: 18-60 Years (HC-HC Diet) (N=7) | Placebo: 18-60 Years (Standard Diet) (N=10) | PF-07258669 6 mg: 18-60 Years (Standard Diet) (N=8) | PF-07258669 20 mg: 18-60 Years (Standard Diet) (N=8) | PF-07258669 60 mg: 18-60 Years (Standard Diet) (N=8) | PF-07258669 125 mg: 18-60 Years (Standard Diet) (N=8) | PF-07258669 180 mg: 18-60 Years (Standard Diet) (N=8) | Placebo: 18-60 Years (HF-HC Diet) (N=12) | PF-07258669 180 mg: 18-60 Years (HF-HC Diet) (N=12) | Placebo: Japanese 18-60 Years (Standard Diet) (N=1) | PF-07258669 180 mg: Japanese 18-60 Years (Standard Diet) (N=5) | Part B Period 1: Midazolam (N=11) | Part B Period 2: PF-07258669 + Midazolam (Day 2) (N=11) | Part B Period 2: PF-07258669 + Midazolam (Day 10) (N=9)
Neurological symptom (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo: 18-60 Years (HC-HC Diet) (N=6) | PF-07258669 2 mg: 18-60 Years (HC-HC Diet) (N=8) | PF-07258669 3 mg: 18-60 Years (HC-HC Diet) (N=8) | PF-07258669 6 mg: 18-60 Years (HC-HC Diet) (N=7) | Placebo: 18-60 Years (Standard Diet) (N=10) | PF-07258669 6 mg: 18-60 Years (Standard Diet) (N=8) | PF-07258669 20 mg: 18-60 Years (Standard Diet) (N=8) | PF-07258669 60 mg: 18-60 Years (Standard Diet) (N=8) | PF-07258669 125 mg: 18-60 Years (Standard Diet) (N=8) | PF-07258669 180 mg: 18-60 Years (Standard Diet) (N=8) | Placebo: 18-60 Years (HF-HC Diet) (N=12) | PF-07258669 180 mg: 18-60 Years (HF-HC Diet) (N=12) | Placebo: Japanese 18-60 Years (Standard Diet) (N=1) | PF-07258669 180 mg: Japanese 18-60 Years (Standard Diet) (N=5) | Part B Period 1: Midazolam (N=11) | Part B Period 2: PF-07258669 + Midazolam (Day 2) (N=11) | Part B Period 2: PF-07258669 + Midazolam (Day 10) (N=9)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nodal arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nodal rhythm (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Delayed light adaptation (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular discomfort (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Change of bowel habit (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Application site irritation (General disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Energy increased (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Feeling cold (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hunger (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thirst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Vaccination site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Food craving (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Poor quality sleep (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 4 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arrhythmia prophylaxis (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vasoconstriction (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Drooling (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Any untoward findings identified on physical and/or neurological examinations, cardiac monitoring and pulse oximeter monitoring conducted during the active collection period were captured as adverse events, if those findings met the definition of an AE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-11-09): https://cdn.clinicaltrials.gov/large-docs/40/NCT05113940/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-04): https://cdn.clinicaltrials.gov/large-docs/40/NCT05113940/SAP_001.pdf